CLINICAL TRIAL: NCT00042133
Title: Socio-economic Status and Age-related Disability in a Biracial Community
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10902-CP-001
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: aging; disability; longitudinal studies; neighborhood factors; socio-economic status; race

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The overall goal of the proposed project is to examine the reasons for the higher levels of disability in older people of lower socio-economic status.

DETAILED DESCRIPTION:
This application is a continuation of an epidemiologic study that investigates the effect of socio-economic disadvantage and neighborhood conditions on disability in older blacks and whites. The proposed project takes place in the context of a population-based, longitudinal study of persons aged 65 years and over who live in a geographically defined, urban, biracial community area in Chicago. During the initial funding period, we have successfully collected yearly disability outcome data, and detailed information on neighborhood conditions using self-report instruments and a systematic neighborhood survey of study area.

The first overall goal of this continuation is to determine the relative contribution and specific nature of the neighborhood conditions that are associated with disability in older adults. The second overall goal is to determine the biological mechanisms through which neighborhood conditions lead to increased disability, focusing specifically on hyperactivity of the hypothalamus-pituitary-adrenal (HPA) axis, via salivary cortisol, and inflammatory processes, via interleukin-6 (IL-6) and C-reactive protein (CRP), obtained from blood samples. To accomplish these goals, we propose to continue yearly collection of disability outcome data and obtain blood samples and salivary cortisol from over 7,000 participants. These data will be integrated with a rich set of existing data on personal characteristics, health conditions, and neighborhood factors to test of series of specific hypotheses related to the overall goals.

Disability is a common and highly prevalent consequence of age-related chronic diseases, and a critical indicator of overall health among older people. Prevention of disability is essential to improve the lives of older people and reduce health care costs. The proposed work will contribute to a better understanding of the specific neighborhood conditions that are associated with increased disability, laying the foundation for more effective policies to prevent disability in future generations of older adults.

ELIGIBILITY:
inclusion criteria: adults aged 65 years and over exclusion criteria: none

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2001-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F. Mendes de Leon, Ph.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States